CLINICAL TRIAL: NCT06372301
Title: Utility of Dobutamine Stress Echocardiography in the Diagnosis of Severe Aortic Stenosis in Patients With Low-flow Low-gradient and Co-exiting Wild-type Transthyretin Amyloid Cardiomyopathy
Brief Title: Dobutamine Stress Echocardiography in LF/LG Aortic Stenosis and Wild-type Transthyretin Amyloid Cardiomyopathy
Acronym: DobAttrAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Professor, DMSc., Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-179-23
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Transthyretin Amyloid Cardiomyopathy; Aortic Stenosis
Keywords: ATTR-CM; wild-type cardiac amyloidosis; aortic stenosis; low-flow low-gradient aortic stenosis; Dobutamine
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Echocardiography, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Co-existing AS and ATTRwt (Experimental): Symptomatic patients with co-existing wild-type transthyretin amyloid cardiomyopathy and low-flow low gradient AS.
  Interventions: Diagnostic Test: Dobutamine stress echocardiography

INTERVENTIONS:
Diagnostic Test: Dobutamine stress echocardiography — Patients will be investigated with dobutamine stress echocardiography (increasing doses of dobutamine infusion and simulatneous echocardiogarphic evaluation) to assess aortic valve area and projected aortic valve area.

SUMMARY:
The goal of this prospective clinical study is improve the diagnosis of Low-flow low-gradient aortic stenosis (LF/LG AS), in patients with co-existing wild-type transthyretin cardiac amyloidosis (ATTRwt). The main question it aims to answer is whether the classic dobutamine-stress echocardiography can be used to determine AS severity in patients with ATTRwt and LF/LG AS This question will be tried to answer by comparing dobutamine stress echocardiography, with the invasively measured aortic valve area (which is considered as the gold standard).

In addition we aim to assess the degree of myocardial fibrosis and amyloid infiltration, assessed by light microscopy and cardiac magnetic resonance (CMRI) and evaluation of myocyte mitochondrial function by high resolution respirometry and their relation to AS severity and hemodynamic response to dobutamine.

DETAILED DESCRIPTION:
Study protocol

A- Baseline assessment: The following will be measured:

* Blood pressure and heart rate.
* ECG.
* Standard echocardiography.
* Dobutamine stress echocardiography.

B- Catheterization laboratory: The participant will be transferred to the catheterization laboratory after about 1.5-hour recovery period after the end of dobutamine stress echocardiography. The following will be done in the following order:

* Right heart catheterization and endomyocardial biopsies.
* Left heart catheterization.
* Dobutamine challenge: Infusion of increasing dobutamine dosages, with simultaneous invasive measurements.
* Removal of left and right heart catheters: The catheters will be removed after 5 minutes recovery after dobutamine challenge.

C- Observation: The participant will then be transferred to our out-patient hospital for observation and the participant is expected to be discharged after 2 hours of observation, if no complications arise.

D- CMRI: All the participants will be evaluated with CMRI for estimation of LV mass, T-1 values, and extracellular volume (ECV). This will be scheduled for a separate visit.

Investigations and procedures

1. Dobutamine Challenges

   Dobutamine challenge will be performed two times at the trial day. The first dobutamine challenge will be performed immediately after the baseline echocardiographic examination. The second dobutamine challenge will be performed no earlier than 2 hours later at the catherization laboratory as described below. Dobutamine, known for its brief half-life of approximately 2 minutes, ensures that its effects diminish rapidly, and the specified two-hour interval guarantees that its influence has subsided.

   A ramp dobutamine infusion will be performed with a stepwise dobutamine dosage increase (dosages: 2,3,5,10,20 ug/kg/min). Dobutamine dosage will only be increased to 40 ug/kg/min in patients with ongoing beta-blocker treatment to ensure an appropriate dobutamine response.

   The first dobutamine challenge with echocardiography: Blood pressure, heart rate, and standard echocardiography images will be obtained before the infusion start, at each infusion stage, and during the recovery period after the infusion is omitted. The projected aortic valve area (AVAproj.) is calculated by using the simplified formula:

   AVAproj =AVArest + " AVApeak- AVArest" /"Qpeak-Qrest" " x (250- Qrest)

   Q is defined as the transvalvular flow rate = SV/Ejection time. SV is calculated by the LVOTVTI x LVOTarea. Ejection time is measured by CW-Doppler of the valve profile.

   The second dobutamine challenge with invasive measurements: This will be performed at the catheterization laboratory after the insertion of right and left heart catheters. There must be a minimum of 2 hours between the two dobutamine challenges. Blood pressure, heart rate, and pressure and flow measurements will be obtained before the infusion start, at each infusion stage, and during the recovery period after the infusion is omitted. AVA will be estimated at rest and at each dobutamine dose level using Gorlin formula.The abovementioned equation for AVAproj. will be also used to calculate AVAproj. from the invasive measurements.
2. Endomyocardial biopsies and biobank Before the right and left heart catheterization are initiated, three endomyocardial biopsies will be taken from the interventricular septum, through the internal jugular vein access (or femoral vein). The first biopsy is for evaluation of mitochondrial function by high resolution respirometry. The other two biopsies are for semi-quantitative evaluation of fibrosis and amyloid infiltration by standard diagnostic light microscopy at the department of pathology at Aarhus University Hospital. Any residual tissue from the first biopsy (to respirometry) will be destroyed after completing the analysis. The biopsies for light microscopy will be prepared, analyzed, and stored in clinical biobank according to the standard clinical practice at the department of pathology.
3. High Resolution Respirometry Biopsies used for high resolution respirometry are analyzed immediately after being taken. High resolution respirometry is performed at the unit of Clinical Research, Department of Cardiology at Aarhus University Hospital. The procedure is standard in the department.
4. Cardiac Magnetic Resonance Imaging (CMRI) CMRI scan will be performed to assess LV mass, fibrosis (assessed as late gadolinium enhancement), ECV assessed using T1-mapping, LV volume, left and right ventricular ejection fraction and strain mapping analysis. Gadolinium-based contrast will not be administered to participants with an estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1,73 m2 due to the risk of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. ATTRwt, diagnosis confirmed by 99mtc-3,3-Diphosphono-1,2-Propanodicarboxylic Acid (DPD) scintigraphy, genetic testing, and/or endomyocardial biopsy.
2. Symptomatic patients (New York Heart Association > class I) treated with loop diuretics.
3. LF/LG AS: Defined as, aortic valve area ≤ 1 cm2 and mean gradient < 40 mmHg, and SVI ≤35 ml/m2.
4. Age ≥ 65 years.
5. Oral and written informed consent.

Exclusion Criteria:

1. Other significant valvular disease.
2. Known severe coronary artery diseases: left main stem stenosis or 3-vessel disease, or recent acute myocardial infarction (< 4 weeks).
3. Contraindications to the use of dobutamine: Known allergy to dobutamine or sulfite, phaeochromocytoma or ventricular tachycardia (VT).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between echocardiography derived projected aortic valve area (AVAproj) and invasively assessed AVAproj under dobutamine infusion. | Evaluated at the end of dobutamine infusion.

SECONDARY OUTCOMES:
Correlation between echocardiography derived AVA and invasively assessed AVA at rest and at different dobutamine infusion levels. | Evaluated at rest, at every dobutamine dose-level, and at the end of infusion.
Increase of SVI, LV ejection fraction and LV-global longitudinal strain of 10 % during maximal dobutamine stimulation. | Evaluated at the end of dobutamine infusion.
Correlation between echo- and invasive measured SVI. | Evaluated at the end of dobutamine infusion.
Degree of myocardial fibrosis, amyloid infiltration and mitochondrial dysfunction and its relation to AS severity and hemodynamic response to dobutamine | CMRI would be performed within a max of 2 months from the trial day.
Reduction of mean pulmonary artery wedge pressure and/or mean pulmonary artery pressure by 10 %. | Evaluated at the end of dobutamine infusion.
Complication rate and symptomatic side effects during dobutamine challenge | Evaluated after couple of days after trial day with dobutamine infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Aarhus, Denmark